CLINICAL TRIAL: NCT02736435
Title: Treatment of Uterine Fibroids With Magnetic Resonance Guided High Intensity Focused Ultrasound
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lengthy delays and inadequate support to proceed.
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-317-07302014
Record Dates: First submitted 2016-03-18; First posted 2016-04-13 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2017-04

CONDITIONS: Uterine Leiomyoma
Keywords: Magnetic Resonance Guided High Intensity Focused Ultrasound; MR-HIFU; Fibroids; Leuprolide Acetate
MeSH Terms: conditions — Myofibroma; Leiomyoma | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fibroid dimension < 8 cm (Experimental): Women with a maximum fibroid dimension less than 8 cm and a total uterine volume less than 900 cc.
  Intervention: Treatment of fibroids with Magnetic Resonance Guided High Intensity Focused Ultrasound.
  Interventions: Device: Magnetic Resonance Guided High Intensity Focused Ultrasound
- Fibroid dimension > 8 cm (Experimental): Women with a maximum fibroid dimension greater than 8 cm or a total uterine volume greater than 900 cc.
  Intervention A: Pre-treated with 11.25mg leuprolide acetate for depot suspension for 3 months to reduce size of fibroids.
  Intervention B: Treatment with Magnetic Resonance Guided High Intensity Focused Ultrasound if fibroids decrease to treatable size of less than 8cm and uterine volume less than 900cc.
  Interventions: Device: Magnetic Resonance Guided High Intensity Focused Ultrasound; Drug: leuprolide acetate for depot suspension

INTERVENTIONS:
Device: Magnetic Resonance Guided High Intensity Focused Ultrasound — Direct treatment of uterine fibroids with MR-HIFU
  Other Names: MR-HIFU
Drug: leuprolide acetate for depot suspension — Treatment of uterine fibroids with leuprolide acetate prior to MR-HIFU
  Other Names: Lupron Depot
  Arms: Fibroid dimension > 8 cm

SUMMARY:
The purpose of this study is to demonstrate the effectiveness of MR-HIFU for the treatment of uterine fibroids in Northwestern Ontario, which is a rural and remote setting.

DETAILED DESCRIPTION:
Uterine fibroids are benign smooth muscle tumours of the muscular wall of the uterus that affect 40 per cent of women. While the majority of fibroids are asymptomatic, fibroids may cause menorrhagia, bulk symptoms (i.e. ureteric obstruction, urinary frequency and urgency, bowel dysfunction), pain and in certain instances infertility.

Magnetic resonance image-guided high-intensity focused ultrasound (MR-HIFU) treatment of fibroids is an established method for symptom alleviation with over 3000 women receiving treatment worldwide. MR-HIFU is a non-invasive, non-surgical procedure that uses ultrasound energy to thermally ablate the fibroid leading to a reduction in bleeding and in the size of uterine fibroids over time. MR-HIFU it is not currently being used for the treatment of symptomatic fibroids in Canada.

The Thunder Bay Regional Research Institute has one of the first clinically available MR-HIFU equipment in Canada. In order to bring this technology into clinical practice, a knowledge translation study is needed to demonstrate that MR-HIFU can treat symptomatic uterine fibroids as successfully in Northwestern Ontario compared to urban centres where all of the clinical trials have been conducted. The ability to screen and follow up women treated with MR-HIFU with ultrasound rather than MRI would allow participants to receive follow up in regional centres in Northwestern Ontario and it would be more cost effective from a health system perspective. In addition, more research is needed to broaden the scope of treatment to include fibroids greater than 8 cm such that more women could benefit from this non-surgical fibroid management option.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 50 years
* Weight <140kg
* Pre or perimenopausal
* Uterine size <24 weeks
* Cervical screen by Pap test: Normal, Low Grade Squamous Intraepithelial Lesion, or Atypical Squamous Cells of Undetermined Significance as per Cancer Care Ontario guidelines
* Transformed symptom severity score ≥40
* Willing to attend all study visits
* Willing to complete evaluation forms
* Willing and able to use reliable contraception;

MR-HIFU Criteria Trial Arm 1:

* Minimum of 50% of fibroid volume accessible for treatment
* Dominant fibroid ≤8 cm
* Uterine volume <900 cc
* Total fibroid treatment volume <250 cc
* No more than 5 fibroids planned for ablation
* Completely non-enhancing fibroids should not be treated

MR-HIFU Criteria Trial Arm 2:

* Minimum of 50% of fibroid volume accessible for treatment
* Dominant fibroid >8 cm or uterine volume >900 cc
* Total fibroid treatment volume <250 cc
* No more than 5 fibroids planned for ablation
* Completely non-enhancing fibroids should not be treated

Exclusion Criteria:

* Other pelvic disease (endometriosis, ovarian tumor, acute pelvic disease, other mass)
* Significant systemic disease even if well controlled
* Positive pregnancy test
* Abnormal uterine bleeding (participant can be included if an endometrial biopsy confirms no hyperplasia or malignancy in the past 6 months)
* Extensive scarring along anterior abdominal wall (>50% of area)
* Surgical clips or scar tissue in the path of the MR-HIFU beam
* MRI contraindicated according to standard operating procedure
* MRI contrast contraindicated (including renal insufficiency)
* Calcifications around or throughout uterine tissues
* Fibroids not quantifiable on MRI
* Highly perfused or brighter than myometrium in T2-weighted MRI fibroids (Type 3 fibroids).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Change in uterine fibroid symptom severity scale | 3, 6, and 12 months
  Assessing change from baseline value

SECONDARY OUTCOMES:
Change in short form McGill pain questionnaire | 24h, 72h, 6week, 3, 6, and 12 month
  Assessing change from baseline value
Change in pictorial blood loss assessment chart | 3, 6, and 12 months
  Assessing change from baseline value
Change in uterine fibroid symptom and health-related quality of life questionnaire | 12 months
  Assessing change from baseline value
Participant use of alternative therapies for treatment of fibroids | 6 weeks, 3, 6, and 12 months
  Questionnaire to assess if participants are selecting to use alternative treatments for relief of symptoms of uterine fibroids.
MR Imaging to assess change in fibroid volume. | 3, 6, and 12 months
  Assessing change from baseline value
MR Imaging to assess change in perfusion. | 3, 6, and 12 months
  Assessing change from baseline value
Ultrasound imaging to assess change in fibroid volume. | 3, 6, and 12 months
  Assessing change from baseline value
Ultrasound imaging to assess change in fibroid perfusion. | 3, 6, and 12 months
  Assessing change from baseline value

OTHER OUTCOMES:
Return to activity within 72 hours of treatment | 72 hours
Change in hemoglobin level | 3, 6, and 12 months
  Assessing change from baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Naana A Jumah, MD DPhil FRCSC, Principal Investigator — Northern Ontario School of Medicine, Thunder Bay Regional Research Institute
Locations (1):
- Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman AJ, Hoffman DI, Comite F, Browneller RW, Miller JD. Treatment of leiomyomata uteri with leuprolide acetate depot: a double-blind, placebo-controlled, multicenter study. The Leuprolide Study Group. Obstet Gynecol. 1991 May;77(5):720-5. PMID 1901638
- [Background] Gizzo S, Saccardi C, Patrelli TS, Ancona E, Noventa M, Fagherazzi S, Mozzanega B, D'Antona D, Nardelli GB. Magnetic resonance-guided focused ultrasound myomectomy: safety, efficacy, subsequent fertility and quality-of-life improvements, a systematic review. Reprod Sci. 2014 Apr;21(4):465-76. doi: 10.1177/1933719113497289. Epub 2013 Jul 18. PMID 23868442
- [Background] Quinn SD, Vedelago J, Gedroyc W, Regan L. Safety and five-year re-intervention following magnetic resonance-guided focused ultrasound (MRgFUS) for uterine fibroids. Eur J Obstet Gynecol Reprod Biol. 2014 Nov;182:247-51. doi: 10.1016/j.ejogrb.2014.09.039. Epub 2014 Oct 6. PMID 25445107
- [Background] Smart OC, Hindley JT, Regan L, Gedroyc WG. Gonadotrophin-releasing hormone and magnetic-resonance-guided ultrasound surgery for uterine leiomyomata. Obstet Gynecol. 2006 Jul;108(1):49-54. doi: 10.1097/01.AOG.0000222381.94325.4f. PMID 16816055
- [Background] Stewart EA, Gostout B, Rabinovici J, Kim HS, Regan L, Tempany CM. Sustained relief of leiomyoma symptoms by using focused ultrasound surgery. Obstet Gynecol. 2007 Aug;110(2 Pt 1):279-87. doi: 10.1097/01.AOG.0000275283.39475.f6. PMID 17666601
- [Background] Thiburce AC, Frulio N, Hocquelet A, Maire F, Salut C, Balageas P, Bouzgarrou M, Hocke C, Trillaud H. Magnetic resonance-guided high-intensity focused ultrasound for uterine fibroids: Mid-term outcomes of 36 patients treated with the Sonalleve system. Int J Hyperthermia. 2015;31(7):764-70. doi: 10.3109/02656736.2015.1063169. Epub 2015 Sep 14. PMID 26367772